CLINICAL TRIAL: NCT00489853
Title: A Multi-centre, Randomised, Double-blind, Cross-over Design Study to Evaluate Efficacy on Exercise Tolerance of Symbicort ®(Budesonide/Formoterol) 320/9μg One Inhalation Twice Daily Compared With Placebo and Oxis® 9μg One Inhalation Twice Daily in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Evaluation of Efficacy on Exercise Tolerance of Symbicort (Budesonide/Formoterol) Compared to Placebo and Oxis in Patients With Severe COPD
Acronym: CODEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5892C00014; Eudract No: 2006-006519-60
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Symbicort then Formoterol then Placebo (Experimental): Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms, 1 inhalation twice daily, then Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily, then Placebo, 1 inhalation twice daily
  Interventions: Drug: budesonide/formoterol Turbuhaler 320/9µg; Drug: formoterol Turbuhaler 9µg; Other: Placebo
- Formoterol then Symbicort then Placebo (Experimental): Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily, then Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms, 1 inhalation twice daily, then Placebo, 1 inhalation twice daily
  Interventions: Drug: budesonide/formoterol Turbuhaler 320/9µg; Drug: formoterol Turbuhaler 9µg; Other: Placebo
- Placebo then Formoterol then Symbicort (Placebo Comparator): Placebo, 1 inhalation twice daily, then Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily, then Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms, 1 inhalation twice daily
  Interventions: Drug: budesonide/formoterol Turbuhaler 320/9µg; Drug: formoterol Turbuhaler 9µg; Other: Placebo

INTERVENTIONS:
Drug: budesonide/formoterol Turbuhaler 320/9µg — Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms
Drug: formoterol Turbuhaler 9µg — Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily
Other: Placebo — Placebo, 1 inhalation twice daily

SUMMARY:
The purpose of this study is to investigate the effect on exercise tolerance, lung function and symptoms after treatment with Symbicort, Oxis or placebo in patients with severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* >=40 years of age
* diagnosed COPD with symptoms >= 2 years
* pre-bronchodilatory FEV1 <=50% of PN

Exclusion Criteria:

* Current respiratory tract disorder other than COPD
* history of asthma or rhinitis
* significant or unstable cardiovascular disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca; Heinrich Worth, MD, Principal Investigator — Akademisches Lehrkrankenhaus der Universität Erlangen-Nürnberg, Germany
Locations (9):
- Germany (8):
  - Research Site, Berlin
  - Research Site, Erfurt
  - Research Site, Fulda
  - Research Site, Fürth
  - Research Site, Geesthacht
  - Research Site, Grobhansdorf
  - Research Site, Leipzig
  - Research Site, Neuruppin
- Research Site, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Worth H, Forster K, Eriksson G, Nihlen U, Peterson S, Magnussen H. Budesonide added to formoterol contributes to improved exercise tolerance in patients with COPD. Respir Med. 2010 Oct;104(10):1450-9. doi: 10.1016/j.rmed.2010.07.006. Epub 2010 Aug 7. PMID 20692140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in 12 centers in Germany and 12 centers in Switzerland.
Pre-assignment Details: Among 137 enrolled patients, 26 patients were not randomised (14 due to violation of inclusion/exclusion criteria, 2 due to adverse events, 1 due to development of study-specific discontinuation criteria, 7 due to voluntary discontinuation, 1 due to lost to follow-up, and 1 due to other reason.)
Period: Treatment Period 1
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 36 | 37 | 38
Completed | 36 | 37 | 38
Not Completed | 0 | 0 | 0
Period: Wash-out Period 1
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 36 | 37 | 38
Completed | 35 | 34 | 32
Not Completed | 1 | 3 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Study-specific discontinuation criteria | 0 | 1 | 4
Period: Treatment Period 2
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 33 | 35 | 33
Completed | 33 | 35 | 33
Not Completed | 0 | 0 | 0
Period: Wash-out Period 2
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 33 | 35 | 33
Completed | 29 | 32 | 31
Not Completed | 4 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Study specific discontinuation criteria | 3 | 2 | 2
Period: Treatment Period 3
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 29 | 30 | 33
Completed | 29 | 29 | 33
Not Completed | 0 | 1 | 0
Not completed — Study specific discontinuation criteria | 0 | 1 | 0
Period: Follow-up Period
Arm/Group | Symbicort Then Formoterol Then Placebo | Formoterol Then Symbicort Then Placebo | Placebo Then Formoterol Then Symbicort
Started | 29 | 29 | 33
Completed | 29 | 29 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Cross over study with 3 Arms. (1)Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms, 1 inhalation twice daily. (2)Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily. (3) Placebo, 1 inhalation twice daily
Arm/Group | Entire Study Population
Number analyzed (Participants) | 111
Age Continuous [Mean (Full Range); unit: Year] | 63.7 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 84

OUTCOME MEASURES:

1. Primary Outcome: Exercise Endurance Time (EET) at 75% of Peak Work Capacity With Cycle Ergometry 1 Hour Post-dose
Description: Treatment means from individual patient data. Patients with only one EET value where excluded since this model, with patient and period as fixed factors, required data from at least two periods.
Time Frame: Single measurement taken1 hour post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Symbicort: Symbicort (budesonide/formoterol) Turbuhaler 320/9 micrograms, 1 inhalation twice daily
- Formoterol: Formoterol Turbuhaler 9 micrograms, 1 inhalation twice daily
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 98 | 99
Seconds | 529 (377) | 441 (292) | 406 (306)

2. Secondary Outcome: Exercise Endurance Time (EET) at 75% of Peak Work Capacity With Cycle Ergometry 6 Hour Post-dose
Description: as for outcome 1
Time Frame: Single measurement taken 6 hours post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 98 | 98
Seconds | 463 (312) | 408 (283) | 388 (306)

3. Secondary Outcome: Forced Expiratory Flow (FEV1) Pre-dose
Description: The mean of the changes for each patient between the pre-dose value at the start of treatment and the pre-dose value after one week of treatment.
Time Frame: Pre-dose at the start of treatment and pre-dose after one week of treatment
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 101
Liters | 0.0830 (0.2480) | 0.0630 (0.2500) | -0.046 (0.1830)

4. Secondary Outcome: Forced Vital Capacity (FVC) Pre-dose
Description: as for outcome 3
Time Frame: Pre-dose at the start of treatment and pre-dose after one week of treatment
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 101
Liters | 0.060 (0.406) | 0.067 (0.407) | -0.094 (0.360)

5. Secondary Outcome: Vital Capacity (VC) Pre-dose (Change From Pre-treatment to Treatment)
Description: as for outcome 3
Time Frame: Pre-dose at the start of treatment and pre-dose after one week of treatment
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 101
Liters | 0.105 (0.3600) | 0.089 (0.370) | -0.083 (0.371)

6. Secondary Outcome: Peak Expiratory Flow (PEF) Before Morning Dose
Description: The change in average value for the run-in or wash-out period to the average value of the subsequent treatment period.
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 97 | 98 | 100
Liters/minute | 1.30 (32.70) | 5.60 (21.50) | -10.00 (27.00)

7. Secondary Outcome: Sleep Score
Description: The change in average value for the run-in or wash-out period to the average value of the subsequent treatment period, with an ordinal scale of 0 (symptoms did not cause a sleep problem) to 4 (did not sleep at all due to symptoms).
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 98 | 99 | 101
Score on Scale | -1.70 (0.47) | -0.03 (0.47) | 0.11 (0.47)

8. Secondary Outcome: Breathlessness Score
Description: The change in average value for the run-in or wash-out period to the average value of the subsequent treatment period, with an ordinal scale of 0 (unaware of any difficulty in breathing) to 4 (almost constant difficulties in breathing). All patients with data from both periods are included.
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 98 | 99 | 101
Score on Scale | -0.12 (0.54) | -0.40 (0.46) | 0.15 (0.49)

9. Secondary Outcome: Chest Tightness Score
Description: The change in average value for the run-in or wash-out period to the average value of the subsequent treatment period, with an ordinal scale of 0 (unaware of any discomfort) to 4 (almost constant discomfort).
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 98 | 99 | 101
Score on a scale | -0.08 (0.46) | -0.02 (0.47) | 0.17 (0.47)

10. Secondary Outcome: Cough Score
Description: The change in average value for the run-in or wash-out period to the average value of the subsequent treatment period, with an ordinal scale of 0 (unaware of coughing) to 4 (never free of need to cough).
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 98 | 99 | 101
Scores on a scale | -0.11 (0.51) | -0.05 (0.50) | 0.10 (0.45)

11. Secondary Outcome: Number of Inhalations of Reliever Medication
Description: The change in average daily use for the run-in or wash-out period to the average daily use of the subsequent treatment period.
Time Frame: Daily diary data entered during the 1-week run-in or wash-out period and the subsequent 1-week treatment period
Measure: Mean (Standard Deviation); unit: Number of inhalations during 24 hours
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 97 | 99 | 101
Number of inhalations during 24 hours | -0.42 (1.51) | -0.36 (1.26) | 0.51 (1.33)

12. Secondary Outcome: Borg CR10 Score Before Exercise Endurance Time (EET) Performed 1 Hour Post-dose
Description: The Borg CR10 Scale consists of 10-point score that the patients pointed to so as to indicate their level of dyspnea before and during exercise testing (where 0 indicates no breathlessness at all and 10 indicates maximum breathlessness. Patients are allowed to assign an even higher number depending on their perceived level of breathlessness).
Time Frame: Single measurement performed at rest prior to exercise endurance test performed 1 hour post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 98 | 98
Scores on a scale | 3.3 (3.2) | 3.4 (3.1) | 3.9 (3.5)

13. Secondary Outcome: Borg CR10 Score After Exercise Endurance Time (EET) Performed 1 Hour Post-dose
Description: The level of breathing discomfort experienced by patients, on a scale of 0 (no breathing discomfort at all) to >10 (absolute maximum breathing discomfort).
Time Frame: Single measurement performed after exercise endurance test performed 1 hour post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 98 | 97
Scores on a scale | 11.5 (2.7) | 11.6 (2.9) | 11.4 (2.9)

14. Secondary Outcome: Borg CR10 Score Before Exercise Endurance Time (EET) Performed 6 Hour Post-dose
Description: as for outcome 13
Time Frame: Single measurement performed at rest prior to exercise endurance test performed 6 hours post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 98 | 98
Scores on a scale | 3.6 (3.2) | 3.4 (3.1) | 3.9 (3.5)

15. Secondary Outcome: Borg CR10 Score After Exercise Endurance Time (EET) Performed 6 Hours Post-dose
Description: The level of breathing discomfort experienced by patients, on a scale of 0 (no breathing discomfort at all) to >10 (absolute maximum breathing discomfort). All patients with data are included.
Time Frame: Single measurement performed after exercise endurance test performed 6 hours post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 94 | 98 | 96
Scores on a scale | 11.5 (2.9) | 11.5 (3.1) | 11.8 (3.1)

16. Secondary Outcome: Inspiratory Capacity (IC) Before Exercise Endurance Time (EET) Performed 1 Hour Postdose
Description: Treatment means from individual participant data.
Time Frame: Single measurement obtained before exercise endurance test performed 1 hour post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 72 | 78 | 70
Liter | 2.06 (0.85) | 2.10 (0.82) | 1.97 (0.72)

17. Secondary Outcome: Inspiratory Capacity (IC) Before Exercise Endurance Time (EET) Performed 6 Hours Post-dose
Description: Treatment means from individual participant data.
Time Frame: Single measurement obtained before exercise endurance test performed 6 hours post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 71 | 78 | 76
Liters | 2.12 (0.79) | 2.12 (0.80) | 1.85 (0.84)

18. Secondary Outcome: Vital Capacity (VC) (Body Plethysmography) Performed Before 1 Hour Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 99 | 102
Liters | 2.75 (0.72) | 2.73 (0.77) | 2.37 (0.66)

19. Secondary Outcome: Inspiratory Capacity (IC) (Body Plethysmography) Performed Before 1 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: Single measurement obtained before exercise endurance test performed 1hour post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 99 | 102
Liters | 2.19 (0.61) | 2.18 (0.70) | 1.91 (0.58)

20. Secondary Outcome: Forced Respiratory Capacity (FRC) (Body Plethysmography) Performed Before 1 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 16
Measure: Median (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 99 | 102
Liters | 5.59 (1.69) | 5.66 (1.61) | 5.79 (1.64)

21. Secondary Outcome: Residual Volume (RV) (Body Plethysmography) Performed Before 1 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 102
Liters | 4.83 (1.59) | 4.94 (1.62) | 5.13 (1.65)

22. Secondary Outcome: Total Lung Capacity (TLC) (Body Plethysmography) Performed Before 1 Hour Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 99 | 102
Liter | 7.58 (1.71) | 7.62 (1.68) | 7.45 (1.76)

23. Secondary Outcome: Specific Airway Resistance (sRaw) (Body Plethysmography) Performed Before 1 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: kilopascal
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 96 | 99 | 101
kilopascal | 2.90 (1.66) | 2.98 (1.81) | 4.22 (2.29)

24. Secondary Outcome: Vital Capacity (VC) (Body Plethysmography) Performed Before 6 Hour Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 100
Liters | 2.69 (0.730) | 2.64 (0.78) | 2.42 (0.71)

25. Secondary Outcome: Inspiratory Capacity (IC) (Body Plethysmography) Performed Before 6 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 100
Liters | 2.14 (0.60) | 2.08 (0.69) | 1.92 (0.66)

26. Secondary Outcome: Forced Respiratory Capacity (FRC) (Body Plethysmography) Performed Before 6 Hours Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 94 | 99 | 99
Liters | 5.47 (1.65) | 5.49 (1.45) | 5.82 (1.88)

27. Secondary Outcome: Residual Volume (RV) (Body Plethysmography) Performed Before 6 Hour Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: Single measurement obtained before exercise endurance test performed 6 hous post-dose at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 94 | 99 | 99
Liters | 4.74 (1.63) | 4.79 (1.52) | 5.19 (1.92)

28. Secondary Outcome: Total Lung Capacity (TLC) (Body Plethysmography) Performed Before 6 Hours Post-dose Exercise Endurance Time (EET)
Description: Treatment means from individual participant data.
Time Frame: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 94 | 99 | 100
Liters | 7.41 (1.68) | 7.37 (1.55) | 7.63 (2.00)

29. Secondary Outcome: Specific Airway Resistance (sRaw) (Body Plethysmography) Performed Before 6 Hours Post-dose EET
Description: Treatment means from individual participant data.
Time Frame: as for outcome 17
Measure: Mean (Standard Deviation); unit: Kilopascals
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 95 | 99 | 100
Kilopascals | 3.06 (1.68) | 3.20 (2.02) | 4.12 (2.54)

30. Secondary Outcome: SGRQ-C (St. George's Respiratory Questionnaire for COPD Patients) Total Score
Description: Score from a questionnaire, with scores ranging form 0 (perfect health) to 100 (worst possible state). Includes all patients with data.
Time Frame: Single measurement taken at the end of each 1-week treatment period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Formoterol | Placebo
Number analyzed (Participants) | 85 | 93 | 91
Scores on a scale | 51.7 (18) | 51.6 (19.2) | 54.5 (18.9)

ADVERSE EVENTS:
Arm/Group | Symbicort | Formoterol | Placebo
Serious Adverse Events (participants affected / at risk) | 2/101 | 1/102 | 1/104
Other Adverse Events (participants affected / at risk) | 4/101 | 3/102 | 6/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=101) | Formoterol (N=102) | Placebo (N=104)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=101) | Formoterol (N=102) | Placebo (N=104)
Chonic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any publication or disclosure, the PI provides AstraZeneca with preliminary data and drafts and with the proposed final manuscript. AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript to review it and may within such time frame require that submission for publication or disclosure be delayed.